CLINICAL TRIAL: NCT02968173
Title: A Prospective, International, Multicenter, Open-Label, Non-Controlled Study of Safety and Effectiveness of Palivizumab, in Children at High Risk of Severe Respiratory Syncytial Virus (RSV) Infection in the Russian Federation and the Republic of Belarus
Brief Title: A Study to Assess the Safety and Effectiveness of Palivizumab Administered to Children at High Risk of Severe Respiratory Syncytial Virus (RSV) Infection in the Russian Federation and the Republic of Belarus
Acronym: Synagis Russia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-539; 2016-000221-39 (EudraCT Number)
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2017-07

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: Bronchopulmonary dysplasia (BPD); RSV hospitalization; Palivizumab; Immunoprophylaxis; Chronic lung disease (CLD) of prematurity
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Congenital chloride diarrhea | interventions — Palivizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Children at High Risk of severe RSV Infection (Experimental): A single IM injection every 30 days beginning at Day 0 for a total of 3-5 injections determined by when in the RSV season a participant was enrolled.
  Interventions: Drug: Palivizumab

INTERVENTIONS:
Drug: Palivizumab — Palivizumab is a humanized immunoglobulin G1 (IgG1) monoclonal antibody directed to an epitope in the A antigenic site of the F (fusion) protein of RSV.
  Other Names: Synagis

SUMMARY:
This is a Phase 3b, prospective, multicenter, open-label, non-controlled study to assess the safety and effectiveness of immunoprophylaxis with the intramuscular (IM) administration of the liquid formulation of palivizumab for the prevention of RSV hospitalizations in infants at high risk (infants born at less than or equal to 35 weeks gestational age and less than or equal to 6 months of age at enrollment; or infants less than or equal to 24 months of age with a diagnosis of chronic lung disease [CLD] of prematurity requiring on-going medical treatment within the previous 6 months or infants less than or equal to 24 months of age with hemodynamically significant congenital heart disease [CHD]).

DETAILED DESCRIPTION:
Participants will receive palivizumab solution for injection at 15 mg/kg by IM injection every 30 days for a minimum of 3 and a maximum of 5 injections given during anticipated periods of RSV risk in the community; the number of doses will depend on the time of enrollment during the RSV season.

ELIGIBILITY:
Inclusion Criteria:

Infants at high risk of severe RSV infection defined as fulfilling at least one of the following:

* Infants born ≤ 35 weeks gestational age AND are ≤ 6 months of age at enrollment
* Infants ≤ 24 months of age at enrollment AND with a diagnosis of bronchopulmonary dysplasia (BPD) (defined as oxygen requirement at a corrected gestational age of 36 weeks) requiring intervention/management (i.e., oxygen, diuretics, bronchodilators, corticosteroids, etc.) anytime within 6 months prior to enrollment
* Infants ≤ 24 months of age at enrollment with hemodynamically significant CHD, either cyanotic or acyanotic, unoperated or partially corrected. Children with acyanotic cardiac lesions must have pulmonary hypertension (≥ 40 mmHg measured pressure in the pulmonary artery [ultrasound acceptable]) or the need for daily medication to manage hemodynamically significant CHD

Exclusion Criteria (main exclusion criteria):

* Hospitalization at the time of enrollment (unless discharge is anticipated within 14 days)
* Mechanical ventilation (including continuous positive airway pressure, CPAP) at the time of enrollment
* Life expectancy less than 6 months
* Unstable cardiac or respiratory status, including cardiac defects so severe that survival is not expected or for which cardiac transplantation is planned or anticipated
* Active respiratory illness, or other acute infection

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Valdes, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Children at High Risk of Severe RSV Infection: A single intramuscular (IM) injection of palivizumab every 30 days beginning at Day 0 for a total of 3-5 injections determined by when in the respiratory syncytial virus (RSV) season a participant was enrolled.
Period: Overall Study
Arm/Group | Children at High Risk of Severe RSV Infection
Started | 50
Completed | 49
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Children at High Risk of Severe RSV Infection: A single IM injection of palivizumab every 30 days beginning at Day 0 for a total of 3-5 injections determined by when in the RSV season a participant was enrolled.
Arm/Group | Children at High Risk of Severe RSV Infection
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: months] | 6.22 (4.428)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With RSV Hospitalization
Description: An RSV hospitalization is defined as either 1) a respiratory/cardiac hospitalization with a positive RSV test, 2) new onset of respiratory/cardiac symptoms in an already hospitalized child, with an objective measure of worsening respiratory/cardiac status and a positive RSV test, or 3) deaths, which can be demonstrated as caused by RSV (by autopsy or clinical history and virologic evidence).
Time Frame: Approximately 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Children at High Risk of Severe RSV Infection
Number analyzed (Participants) | 50
percentage of participants | 0.0 [0.0 to 7.1]

2. Secondary Outcome: Total Number of RSV-Hospitalization Days
Time Frame: Approximately 6 months
Population: All secondary outcome measures were dependent on RSV hospitalization. Since no participants experienced an RSV hospitalization during the study, an evaluation of these outcome measures was not applicable.
Arm/Group | Children at High Risk of Severe RSV Infection
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants Who Received Supplemental Oxygen While Hospitalized
Description: Increased supplemental oxygen is defined as a new requirement or an increase in supplemental oxygen from prior to the onset of cardiac/respiratory symptoms.
Time Frame: Approximately 6 months
Population: as for outcome 2
Arm/Group | Children at High Risk of Severe RSV Infection
Number analyzed (Participants) | 0

4. Secondary Outcome: Total RSV-hospitalization Days With Increased Supplemental Oxygen Requirement
Description: as for outcome 3
Time Frame: Approximately 6 months
Population: as for outcome 2
Arm/Group | Children at High Risk of Severe RSV Infection
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Intensive Care Unit (ICU) Admissions During RSV-hospitalization
Time Frame: Approximately 6 months
Population: as for outcome 2
Arm/Group | Children at High Risk of Severe RSV Infection
Number analyzed (Participants) | 0

6. Secondary Outcome: Total Days of RSV-ICU Stay
Time Frame: Approximately 6 months
Population: as for outcome 2
Arm/Group | Children at High Risk of Severe RSV Infection
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of Participants Who Received Mechanical Ventilation
Time Frame: Approximately 6 months
Population: as for outcome 2
Arm/Group | Children at High Risk of Severe RSV Infection
Number analyzed (Participants) | 0

8. Secondary Outcome: Total Days of Mechanical Ventilation During RSV-hospitalization
Time Frame: Approximately 6 months
Population: as for outcome 2
Arm/Group | Children at High Risk of Severe RSV Infection
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose of study treatment through the last prophylaxis visit (up to Day 120 [±5 days]) + 30 days (+5 days) and 100 days (+5 days)
Groups:
- PALIVIZUMAB TEAE Within 30 Days: A single IM injection of palivizumab every 30 days beginning at Day 0 for a total of 3-5 injections determined by when in the RSV season a participant was enrolled.
  Treatment-emergent adverse events (TEAEs) are defined as those that began after the first dose of study drug but within 30 days (+ 30 day assessment period) after the last dose of study drug.
- PALIVIZUMAB TEAE Within 100 Days: A single IM injection of palivizumab every 30 days beginning at Day 0 for a total of 3-5 injections determined by when in the RSV season a participant was enrolled.
  TEAEs are defined as those that began after the first dose of study drug but within 100 days (+ 100 day assessment period) after the last dose of study drug.
Arm/Group | PALIVIZUMAB TEAE Within 30 Days | PALIVIZUMAB TEAE Within 100 Days
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 6/50 | 6/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PALIVIZUMAB TEAE Within 30 Days (N=50) | PALIVIZUMAB TEAE Within 100 Days (N=50)
Tachycardia paroxysmal (Cardiac disorders) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 1
Bronchitis viral (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT02968173/SAP_000.pdf
  • Study Protocol (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT02968173/Prot_001.pdf